CLINICAL TRIAL: NCT06342648
Title: Comparison Between Intracutaneous Sterile Water and Diclofenac Sodium Injections in Renal Colic: A Randomized Controlled Clinical Trial
Brief Title: Intracutaneous Sterile Water and Diclofenac Sodium Injections in Renal Colic
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Principal Investigator, Abdelrhman Alshawadfy, Clinical Professor Suez Canal University Faculty of Medicine, Suez Canal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Cutaneous water in renal colic
Record Dates: First submitted 2024-03-19; First posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Renal Colic
MeSH Terms: conditions — Renal Colic | interventions — Diclofenac

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intracutaneous sterile water injection (ISWI) (Active Comparator): Sterile water will be intramuscularly injected in the intracutaneous sterile water injection (ISWI) group (Group I) in a plane parallel to the posterior midline, adhering to a predetermined injection pattern from the level of the iliac crest to the last rib.
  Interventions: Drug: Sterile Water Injection
- Intramuscular diclofenac sodium injection (DIC) (Active Comparator): Diclofenac sodium injection intramuscularly (Group II): Diclofenac sodium injection intramuscularly (75 mg) will be given to 285 patients in total.
  Interventions: Drug: Diclofenac Sodium injection

INTERVENTIONS:
Drug: Sterile Water Injection — Injection of intracutaneous sterile water
  Arms: Intracutaneous sterile water injection (ISWI)
Drug: Diclofenac Sodium injection — Injection of intramuscular diclofenac sodium
  Arms: Intramuscular diclofenac sodium injection (DIC)

SUMMARY:
Renal colic is a serious and excruciatingly painful condition that frequently presents itself in the emergency department. In this trial, patients with renal colic who have received intramuscular diclofenac sodium injection or intracutaneous sterile water injection will have their Visual Analogue Scale (VAS) measured and compared.

DETAILED DESCRIPTION:
Renal colic affects over 12% of the global population at some point in their lives, and recurrence rates are 50%. Renal colic affects approximately 1.2 million people annually and is the reason for 1% of emergency department visits and hospital stays. Urinary tract obstruction caused by calculi is the most common cause of renal colic occurrence. The sudden onset of colicky pain that begins in the flank and radiates to the groin is the classic clinical feature of a ureteric colic. Most people agree that this pain is the worst that humans have ever felt. Renal colic pain can be effectively managed with a variety of pharmacologic treatments, including nonsteroidal anti-inflammatory drugs (NSAIDs), opioid analgesics, antispasmodics, and antidiuretic hormones. However, the best analgesic regimen has not yet been identified. In patients with renal colic, intravenous (IV) injections of analgesics-either opioids or NSAIDs-remain standard clinical procedures for managing pain. While there have been reports of success with IV administration of these medications, side effects and availability are typically problematic, particularly in private clinics or with opioid abuse. Furthermore, because NSAIDs may reduce renal blood flow and obstruct the kidney's autoregulatory response to obstruction, preexisting renal disease may exacerbate renal failure. The majority of doctors are also uncomfortable using these medications because of their side effects, which include hypotension, respiratory depression, dizziness, nausea, vomiting, narcotic dependence, sedation, and lightheadedness. Therefore, it would appear that using alternate treatments to manage renal colic pain is inevitable. In this trial, the investigators will compare the Visual Analogue Scale (VAS) in patients with renal colic after being managed with intracutaneous sterile water injection and intramuscular diclofenac sodium injection.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18 and 65.
* Patients with renal colic at the emergency department of the 30 June Center for Urology and Nephrology, Ismailia, Egypt.

Exclusion Criteria:

* Cardiovascular diseases.
* Renal, and hepatic dysfunction.
* Hypersensitivity to any of the used drugs.
* Addiction or chronic use of opioids.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 570 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | For 45 minutes, the VAS will be measured three times, at 15, 30, and 45 minutes of the procedure.
  Comparing the Visual Analogue Scale (VAS) between patients who had intramuscular diclofenac sodium injection and intracutaneous sterile water injection for the treatment of renal colic. One of the pain rating instruments that Hayes and Patterson used for the first time was the Visual Analogue Scale (VAS), introduced in 1921. A straight line represents the visual analog scale for pain, with zero representing no pain and ten representing the worst possible pain. A patient indicates on the line the location of the point that corresponds to their level of pain.